CLINICAL TRIAL: NCT03835546
Title: Observational Prospective Trial to Investigate the Impact of Antiretroviral Therapy Initiation With Integrase Strand Transfer Inhibitors on Brain Outcomes:The ARBRE Study:Impact of AntiRetroviral Therapy With INSTI on BRain outcomEs (ARBRE) According to the Time of Therapy Initation
Brief Title: Study to Assess the ART Impact on the Brain Outcomes. The ARBRE Study
Acronym: ARBRE
Status: Completed | Type: Observational
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: Institut de Diagnostic per la Imatge (Other); Institut d'Investigació Biomèdica de Bellvitge (Other); Consorci Sanitari de Terrassa (Other); BCN Checkpoint (Industry); Germans Trias i Pujol Hospital (Other); IrsiCaixa (Other)
Responsible Party: Sponsor
Other Study IDs: FLS-ANT-2015-01
Record Dates: First submitted 2018-09-25; First posted 2019-02-08 (Actual); Results first posted 2020-06-01 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: HIV-1 Infection; Cognitive Impairment
Keywords: Brain; HIV-1 Infection
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Early treated patients: Patients with confirmed HIV-1 infection attended in the HIV Unit of the Hospital Universitari Germans Trias i Pujol who initiated therapy presenting recent HIV-1 infection. Recent HIV-1 infection was defined as having a positive plasma viral load and/or p24 antigen with a negative ELISA or having a positive ELISA and undetermined Western-Blot, or having a positive ELISA and absence of p31 antigen in a positive Western-Blot, or seroconversion ELISA in less than 3 months.
- Regularly treated patients: Patients with confirmed HIV-1 infection attended in the HIV Unit of the Hospital Universitari Germans Trias i Pujol who initiated therapy, did not fulfil the criteria for recent HIV-1 infection, and had an estimated time >6 months reported by the patient and/or by the responsible physician since HIV transmission.
- Seronegative volunteers: HIV-uninfected volunteers, matched to age, sex, and educational level with groups A and B.

SUMMARY:
The ARBRE Study is an observational prospective trial aimed at investigating the impact of the therapy initiation with INTIs on brain outcomes according to the time of therapy initiation. Three study arms are considered: 1) Early treated HIV-1 infected patients (<3 months since estimated date of infection), 2) Regularly treated HIV-1 infected patients (>6 months since estimated date of infection), 3) Matched seronegative control group. Study assessments will be performed at baseline, 1 month and 12 months. Study assessments will comprise comprehensive evaluation of brain outcomes. They will include cognitive functioning, neuroimaging parameters, and functional outcomes.

DETAILED DESCRIPTION:
Randomized patients will receive LA CAB+RPV administration in the hospital (standard of care) or out-of- hospital administration every 2 months (M2, M4, M6, M8,M10, M12). Medical visits, rutinary blood tests and pharmacy visits at the hospital of reference will take place every 6 months- at baseline, M1 (if patient has not previously receiving LA CAB+RPV), M6 and M12.

ELIGIBILITY:
The study criteria for participation in the study will be the following:

Inclusion Criteria:

* Age 18-65 years old
* Voluntary participation.
* Signed written consent.
* Confirmed HIV-1 infection (for arms A and B).
* Intention to initiate therapy with cART containing an INSTI. Specifically, the regimen included raltegravir, elvitegravir or dolutegravir.

Exclusion Criteria:

* Prior diagnosis of opportunistic infection involving CNS.
* Current diagnosis of psychiatric disorder.
* Current or past diagnosis of neurologic disease.
* Inability to develop any of the tasks required for the study.
* Pregnancy.
* History of suboptimal adherence (for arms A and B).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV patients early treated HIV chronically patients non HIV participants
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-10-26 (Actual); Primary Completion 2016-12-23 (Actual); Study Completion 2018-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose A. Muñoz-Moreno, Principal Investigator — Lluita contra la Sida Foundation

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Early Treated Patients | Regularly Treated Patients | Seronegative Volunteers
Started | 15 | 15 | 15
Completed | 12 | 15 | 15
Not Completed | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Treated Patients | Regularly Treated Patients | Seronegative Volunteers | Total
Number analyzed (Participants) | 12 | 15 | 15 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 15 | 15 | 42
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (10) | 31 (9) | 32 (10) | 32 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 12 | 15 | 15 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 15 | 15 | 42
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 12 | 15 | 15 | 42

OUTCOME MEASURES:

1. Primary Outcome: Change in Global Cognitive Functioning
Description: The measure used will be NPZ-12 (NeuroPsychological Z-12). Minimum value: -5 Maximum value: +5. Mean: 0. Lower score will represent worse global cognitive functioning; higher score will represent better global cognitive functioning.
Time Frame: From Baseline to Week 48
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early Treated Patients | Regularly Treated Patients | Seronegative Volunteers
Number analyzed (Participants) | 12 | 15 | 15
score on a scale | 0.08 (0.26) | 0.31 (0.28) | 0.25 (0.19)

2. Secondary Outcome: Change in Neuropsychiatric Symptoms
Description: The measure used will be a checklist of symptoms involving the central nervous system. Minimum value: 0; Maximum value: 140. Lower score will represent better neuropsychiatric status; higher score will represent worse neuropsychiatric status.
Time Frame: From Baseline to Week 48
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early Treated Patients | Regularly Treated Patients | Seronegative Volunteers
Number analyzed (Participants) | 12 | 15 | 15
score on a scale | -2.90 (8.76) | 0.33 (7.58) | 0.30 (5.77)

3. Secondary Outcome: Change in Daily Living Functioning
Description: Daily living functioning will be measured by a self-reported scale indicating daily living areas impaired. Minimum score: 0; Maximum score: 13. A lower score will represent better daily functioning; a higher score will represent worse daily functioning.
Time Frame: From Baseline to Week 48
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early Treated Patients | Regularly Treated Patients | Seronegative Volunteers
Number analyzed (Participants) | 12 | 15 | 15
score on a scale | 0.54 (1.69) | 0.33 (2.01) | 0.30 (0.82)

4. Secondary Outcome: Change in Depressive Symptoms
Description: Depressive symptoms will be measured by a self-reported scale that will assess depressive symptoms. Minimum score: 0; Maximum score: 21. A lower score will represent better depressive status; a higher score will represent worse depressive status.
Time Frame: From baseline to week 48
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early Treated Patients | Regularly Treated Patients | Seronegative Volunteers
Number analyzed (Participants) | 12 | 15 | 15
score on a scale | -3.55 (2.58) | -0.50 (3.84) | -0.60 (1.43)

5. Secondary Outcome: Change in Anxiety Symptoms
Description: Anxiety symptoms will be measured by a self-reported scale that will assess anxiety symptoms. Minimum score: 0; Maximum score: 21. A lower score will represent better anxiety status; a higher score will represent worse anxiety status.
Time Frame: From Baseline to Week 48
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early Treated Patients | Regularly Treated Patients | Seronegative Volunteers
Number analyzed (Participants) | 12 | 15 | 15
score on a scale | -5.18 (3.46) | -2.00 (2.93) | -1.30 (2.49)

6. Secondary Outcome: Change in Daily Perceived Stress
Description: Perceived stress will be measured by a self-reported scale that will assess daily symptoms of perceived stress. Minimum score: 0; Maximum score: 40. A lower score will represent better perceived stress status; a higher score will represent worse perceived stress status.
Time Frame: From baseline to week 48
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early Treated Patients | Regularly Treated Patients | Seronegative Volunteers
Number analyzed (Participants) | 12 | 15 | 15
score on a scale | -7.55 (3.88) | -6.50 (9.24) | 1.40 (4.72)

7. Secondary Outcome: Change in Quality of Life
Description: Quality of life will be measured by a self-reported scale that will assess global quality of life. Minimum score: 1; Maximum score: 4. A lower score will represent worse quality of life; a higher score will represent better quality of life.
Time Frame: From Baseline to Week 48
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early Treated Patients | Regularly Treated Patients | Seronegative Volunteers
Number analyzed (Participants) | 12 | 15 | 15
score on a scale | 0.18 (0.40) | 0.08 (0.51) | 0.10 (0.73)

8. Secondary Outcome: Change in Neuroimaging Markers
Description: Neuroimaging markers will be assessed by 3T magnetic resonance imaging (MRI). The specific markers will be caudate nucleus, ventral striatum/nucleus accumbens, putamen, pallidum, thalamus, dorsomedial, dorsolateral, cingulate, ventromedial, medial orbitofrontal, and lateral orbitofrontal cortex. The outcome will be based on change in any of them.
Time Frame: From Baseline to Week 48
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From Baseline to week 48
Arm/Group | Early Treated Patients | Regularly Treated Patients | Seronegative Volunteers
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/12 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes